CLINICAL TRIAL: NCT06839404
Title: Pharmacodynamic Analysis of the HaemOdynamic Effects of a Standard Fluid BolUS - the PHOEBUS Study
Brief Title: Pharmacodynamic Analysis of the HaemOdynamic Effects of a Standard Fluid BolUS
Acronym: PHOEBUS
Status: Recruiting | Type: Observational
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Christopher Lai, Doctor, Bicetre Hospital
Other Study IDs: PHOEBUS study; SRLF 22-033 (Other: Ethics committee of the French Intensive Care Society)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: fluid challenge — Fluid bolus of 500 mL of crystalloids given at a constant rate between 10 and 15 minutes

SUMMARY:
When the flow of blood ejected by the heart drops significantly, that is to say when there is "shock", one of the first treatments undertaken is often volume expansion. This treatment consists of injecting a liquid intravenously, generally in the form of a bolus, that is to say a dose of solute administered all at once, of 250 to 500 mL of fluid over approximately 10 to 30 minutes. The injected fluid expands the blood volume and fills the heart pump, in order to increase the flow it ejects.

However, this treatment poses two problems. First, it is only inconsistently effective. It is possible that of the 250-500 mL of fluid administered in the standard way, only a part is effective, whereas, as the effectiveness decreases during the infusion, the rest does not increase cardiac output significantly.

However, the average part of the total volume that is ineffective on a large population of patients is not well known.

Second, the effects of volume expansion on cardiac output decrease rapidly after the end of administration. However, the average duration of effectiveness of a 250-500 mL fluid bolus, and the factors that influence this duration of effectiveness, are not well determined.

The main objective of this research is to measure, among the volume of a fluid bolus, which part does not significantly increase cardiac output. The secondary objective is to measure the average time of effectiveness after the end of the infusion and the factors that influence it.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Hospitalisation in intensive care
* Haemodynamic monitoring already in place with a pulse wave contour analysis-derived estimation of cardiac output (either calibrated or uncalibrated)
* Decision taken by the clinicians in charge of the patient to perform volume expansion by intravenous infusion of a 6 mL/kg crystalloid bolus

Exclusion Criteria:

* Pregnancy
* Refusal to participate by relatives of the patient or the patient himself
* Other therapeutic modification during volume expansion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care unit and with shock for whom a fluid challenge is administered
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To measure, during the administration of a fluid bolus in order to perform volume expansion, the volume of fluid which causes an increase in cardiac output of less than 15%. | During the fluid bolus administration (<15min)
  We will measure, among the volume administered (500mL), the proportion of infused volume which allowed an increase in cardiac output ≥15% compared to the baseline value. This baseline value will be defined by the average measured over the minute preceding the start of the fluid infusion

SECONDARY OUTCOMES:
The maximum amplitude of the change induced by volume expansion in cardiac output, mean arterial pressure and central venous pressure | During the fluid bolus administration (<15min)
  The maximum amplitude, expressed as an absolute value and as a percentage of the baseline value, as defined above, of the change induced by volume expansion in cardiac output, mean arterial pressure and central venous pressure
The delay at which this maximum effect appears in terms of cardiac output, mean arterial pressure and central venous pressure | During the fluid bolus administration (<15min)
The time following the end of the infusion from which the cardiac output becomes ≤5% of the baseline value | A period of 120 minutes following the fluid infusion
The factors that influence these pharmacokinetic variables will be determined | During the study period (during fluid administration and the period of 120 minutes following the infusion)

CONTACTS AND LOCATIONS:
Locations (1):
- Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR